CLINICAL TRIAL: NCT03114969
Title: An Open-label, Low Interventional Clinical Study Investigating Error Rates (Critical and Overall) Prior to Any Retraining in Correct Use of the ELLIPTA Dry Powder Inhaler (DPI) Compared to Other DPIs Including; DISKUS, Turbuhaler, HandiHaler and Breezhaler as a Monotherapy or in Combination, in Adult Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Comparative Study of Error Rates Between ELLIPTA® Dry Powder Inhaler (DPI) and Other DPIs
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 204981
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Results first posted 2019-06-10 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Overall error; Error rate; Critical error; COPD; ELLIPTA; Dry powder inhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Subjects using RELVAR ELLIPTA: Subjects with a fixed dose combination of inhaled corticosteroids/ long-acting beta agonists (ICS/LABA) via a single DPI of RELVAR ELLIPTA for treatment of COPD will be included.
  Interventions: Device: Relvar ELLIPTA
- Subjects using SYMBICORT TURBUHALER: Subjects with a fixed dose combination of ICS/LABA via a single DPI of SYMBICORT TURBUHALER for treatment of COPD will be included.
  Interventions: Device: Symbicort TURBUHALER
- Subjects using SERETIDE DISKUS: Subjects with a fixed dose combination of ICS/LABA via a single DPI of SERETIDE DISKUS for treatment of COPD will be included.
  Interventions: Device: Seretide DISKUS
- Subjects using SPIRIVA HANDIHALER: Subjects with a fixed dose monotherapy of long-acting muscarinic antagonists (LAMA) via a single DPI of SPIRIVA HANDIHALER for treatment of COPD will be included.
  Interventions: Device: Spiriva HANDIHALER
- Subjects using INCRUSE ELLIPTA or ANORO ELLIPTA: Subjects with a fixed dose monotherapy of LAMA via a single DPI of INCRUSE ELLIPTA or subjects taking a fixed dose combination of LAMA/LABA via a single DPI of ANORO ELLIPTA for treatment of COPD will be included.
  Interventions: Device: Incruse ELLIPTA; Device: Anoro ELLIPTA
- Subjects using SEEBRI BREEZHALER or ULTIBRO BREEZHALER: Subjects with a fixed dose monotherapy of LAMA via a single DPI of SEEBRI BREEZHALER or subjects taking a fixed dose combination of LAMA/LABA via a single DPI of ULTIBRO BREEZHALER for treatment of COPD will be included.
  Interventions: Device: BREEZHALER
- Subjects using RELVAR ELLIPTA with HANDIHALER/ INCRUSE ELLIPTA: Subjects with a fixed dose combination of ICS/LABA via RELVAR ELLIPTA along with a fixed dose of LAMA via SPIRIVA HANDIHALER or INCRUSE ELLIPTA will be included.
  Interventions: Device: Relvar ELLIPTA; Device: Spiriva HANDIHALER; Device: Incruse ELLIPTA
- Subjects using TURBUHALER with HANDIHALER/INCRUSE ELLIPTA: Subjects with a fixed dose combination of ICS/LABA via SYMBICORT TURBUHALER along with a fixed dose of LAMA via SPIRIVA HANDIHALER or INCRUSE ELLIPTA will be included.
  Interventions: Device: Symbicort TURBUHALER; Device: Spiriva HANDIHALER; Device: Incruse ELLIPTA
- Subjects using DISKUS with HANDIHALER/INCRUSE ELLIPTA: Subjects with a fixed dose combination of ICS/LABA via SERETIDE DISKUS along with a fixed dose of LAMA via SPIRIVA HANDIHALER or INCRUSE ELLIPTA will be included.
  Interventions: Device: Seretide DISKUS; Device: Spiriva HANDIHALER; Device: Incruse ELLIPTA

INTERVENTIONS:
Device: Relvar ELLIPTA — ELLIPTA inhaler containing Relvar will be used by subjects as their maintenance treatment to control COPD.
  Groups: Subjects using RELVAR ELLIPTA; Subjects using RELVAR ELLIPTA with HANDIHALER/ INCRUSE ELLIPTA
Device: Symbicort TURBUHALER — TURBUHALER inhaler containing Symbicort will be used by subjects as their maintenance treatment to control COPD.
  Groups: Subjects using SYMBICORT TURBUHALER; Subjects using TURBUHALER with HANDIHALER/INCRUSE ELLIPTA
Device: Seretide DISKUS — DISKUS inhaler containing Seretide will be used by subjects as their maintenance treatment to control COPD.
  Groups: Subjects using DISKUS with HANDIHALER/INCRUSE ELLIPTA; Subjects using SERETIDE DISKUS
Device: Spiriva HANDIHALER — HANDIHALER inhaler containing Spiriva will be used by subjects as their maintenance treatment to control COPD.
  Groups: Subjects using DISKUS with HANDIHALER/INCRUSE ELLIPTA; Subjects using RELVAR ELLIPTA with HANDIHALER/ INCRUSE ELLIPTA; Subjects using SPIRIVA HANDIHALER; Subjects using TURBUHALER with HANDIHALER/INCRUSE ELLIPTA
Device: BREEZHALER — BREEZHALER inhaler containing either Seebri or Ultibro will be used by subjects as their maintenance treatment to control COPD.
  Groups: Subjects using SEEBRI BREEZHALER or ULTIBRO BREEZHALER
Device: Incruse ELLIPTA — ELLIPTA inhaler containing Incruse will be used by subjects as their maintenance treatment to control COPD.
  Groups: Subjects using DISKUS with HANDIHALER/INCRUSE ELLIPTA; Subjects using INCRUSE ELLIPTA or ANORO ELLIPTA; Subjects using RELVAR ELLIPTA with HANDIHALER/ INCRUSE ELLIPTA; Subjects using TURBUHALER with HANDIHALER/INCRUSE ELLIPTA
Device: Anoro ELLIPTA — ELLIPTA inhaler containing Anoro will be used by subjects as their maintenance treatment to control COPD.
  Groups: Subjects using INCRUSE ELLIPTA or ANORO ELLIPTA

SUMMARY:
For effective drug delivery using inhalation route, it is important to use the inhalers correctly. This open-label study will evaluate the error rates during the use of ELLIPTA DPI, alone or in combination, in comparison with other DPIs. The study aims to provide clinical evidence in subjects with COPD that the reduced number of steps required to use the ELLIPTA DPI could result in fewer errors made by subjects, and therefore a more consistent treatment. Approximately 450 subjects prescribed with either of RELVAR® ELLIPTA, ANORO® ELLIPTA, INCRUSE® ELLIPTA, SYMBICORT® TURBUHALER®, SERETIDE® DISKUS®, SPIRIVA® HANDIHALER®, ULTIBRO® BREEZHALER® or SEEBRI® BREEZHALER will be included in the study and will have 2 clinical visits. At Visit 1, subjects will take their maintenance DPIs and the critical and overall errors made by subjects will be assessed. After the assessment, subjects will be instructed on correct use or informed of their correct use of their DPIs. The total duration of the study is approximately 6 weeks. ELLIPTA, SERETIDE and DISKUS are registered trademarks of the GSK group of companies. SYMBICORT and TURBUHALER are registered trademarks of the AstraZeneca group of companies. SPIRIVA and HANDIHALER are registered trademarks of Boehringer Ingelheim Pharmaceuticals. ULTIBRO, BREEZHALER and SEEBRI are registered trademarks of the Novartis group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented Physician's diagnosis of COPD, and currently receiving maintenance therapy.
* Aged >=40 years of age at inclusion.
* Using one of the maintenance therapies of interest for at least 3 months prior to inclusion on the study.
* Males or females.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Asthma: Subjects with a current diagnosis of asthma. Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD.
* Drug/alcohol abuse: Subjects with a known or suspected alcohol or drug abuse history at screening (Visit 0) that in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirement.
* Investigational product: Subjects who have received an investigational drug and/or medical device within 30 days of entry into this study (Screening/Visit 1), or within five half-lives of the investigational drug, whichever is longer.
* Investigational product: Subjects who have been trained during participation in any device study in the 6 months prior to entry into this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic obstructive pulmonary disease and uses a dry powder inhaler
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Netherlands (9):
  - GSK Investigational Site, Beek
  - GSK Investigational Site, Beek en Donk
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Kloosterhaar
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Zutphen
- United Kingdom (3):
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, London
  - GSK Investigational Site, Sidcup, Kent

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20591

REFERENCES:
- [Background] Collier DJ, Wielders P, van der Palen J, Heyes L, Midwinter D, Collison K, Preece A, Barnes N, Sharma R. Critical Error Frequency and the Impact of Training with Inhalers Commonly used for Maintenance Treatment in Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2020 Jun 9;15:1301-1313. doi: 10.2147/COPD.S224209. eCollection 2020. PMID 32606640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study investigating error rates for ELLIPTA dry powder inhaler (DPI), alone or in combination when compared to other DPIs (DISKUS, Turbuhaler, HandiHaler and Breezhaler) and combinations of these, as prescribed to chronic obstructive pulmonary disease (COPD) participants, prior to any retraining in correct use.
Pre-assignment Details: A total of 461 participants were screened of which 11 failed screening and 450 participants were enrolled. The study was conducted in two countries-Netherlands and the United Kingdom.
Groups:
- Relvar Ellipta: Participants prescribed a fixed dose combination of inhaled corticosteroid/long-acting beta agonist (ICS/LABA) via Relvar Ellipta for treatment of COPD were included. Participants were assessed for errors while using Relvar Ellipta prior to retraining on the correct use of Ellipta DPI at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of Relvar Ellipta within 6 weeks at Visit 2.
- Symbicort Turbuhaler: Participants prescribed a fixed dose combination of ICS/LABA via Symbicort Turbuhaler for treatment of COPD were included. Participants were assessed for errors while using Symbicort Turbuhaler prior to retraining on the correct use of Turbuhaler at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of Symbicort Turbuhaler within 6 weeks at Visit 2.
- Seretide Diskus: Participants prescribed a fixed dose combination of ICS/LABA via Seretide Diskus for treatment of COPD were included. Participants were assessed for errors while using Seretide Diskus prior to retraining on the correct use of Diskus at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of Seretide Diskus within 6 weeks at Visit 2.
- Spiriva Handihaler: Participants prescribed a fixed dose of long-acting muscarinic antagonist (LAMA) via Spiriva Handihaler for treatment of COPD were included. Participants were assessed for errors while using Spiriva Handihaler prior to retraining on the correct use of Handihaler at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of Spiriva Handihaler within 6 weeks at Visit 2.
- Incruse/Anoro Ellipta: Participants prescribed a fixed dose of LAMA via Incruse Ellipta or participants taking a fixed dose combination of LAMA/LABA via Anoro Ellipta for treatment of COPD were included. Participants were assessed for errors while using Incruse/Anoro Ellipta prior to retraining on the correct use of DPI at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of Incruse/Anoro Ellipta within 6 weeks at Visit 2.
- Ultibro/Seebri Breezhaler: Participants prescribed a fixed dose of LAMA via Seebri Breezehaler or participants taking a fixed dose combination of LAMA/LABA via a single DPI of Ultibro Breezehaler for treatment of COPD were included. Participants were assessed for errors while using Ultibro/Seebri Breezehaler prior to retraining on the correct use of DPI at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of Ultibro/Seebri Breezehaler within 6 weeks at Visit 2.
- Relvar Ellipta+LAMA: Participants prescribed a fixed dose combination of ICS/LABA via Relvar Ellipta along with a fixed dose of LAMA via Spiriva Handihaler or Incruse Ellipta were included. Participants were assessed for errors while using combination DPI prior to retraining on the correct use of DPI at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of combination DPI within 6 weeks at Visit 2.
- Symbicort Turbuhaler+LAMA: Participants prescribed a fixed dose combination of ICS/LABA via Symbicort Turbuhaler along with a fixed dose of LAMA via Spiriva Handihaler or Incruse Ellipta were included. Participants were assessed for errors while using combination DPI prior to retraining on the correct use of DPI at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of combination DPI within 6 weeks at Visit 2.
- Seretide Diskus+LAMA: Participants prescribed a fixed dose combination of ICS/LABA via Seretide Diskus along with a fixed dose of LAMA via Spiriva Handihaler or Incruse Ellipta were included. Participants were assessed for errors while using combination DPI prior to retraining on the correct use of DPI at Visit 1 (Day 1). The participants were retrained on inhaler use following which they were reassessed for errors during use of combination DPI within 6 weeks at Visit 2.
Period: Overall Study
Arm/Group | Relvar Ellipta | Symbicort Turbuhaler | Seretide Diskus | Spiriva Handihaler | Incruse/Anoro Ellipta | Ultibro/Seebri Breezhaler | Relvar Ellipta+LAMA | Symbicort Turbuhaler+LAMA | Seretide Diskus+LAMA
Started | 50 | 50 | 50 | 50 | 51 | 49 | 50 | 50 | 50
Completed | 50 | 50 | 46 | 48 | 51 | 48 | 49 | 50 | 48
Not Completed | 0 | 0 | 4 | 2 | 0 | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relvar Ellipta | Symbicort Turbuhaler | Seretide Diskus | Spiriva Handihaler | Incruse/Anoro Ellipta | Ultibro/Seebri Breezhaler | Relvar Ellipta+LAMA | Symbicort Turbuhaler+LAMA | Seretide Diskus+LAMA | Total
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 51 | 49 | 50 | 50 | 50 | 450
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (10.24) | 65.2 (11.43) | 68.7 (10.67) | 69.5 (9.95) | 66.8 (8.93) | 67.7 (10.01) | 66.6 (8.44) | 67.5 (8.21) | 68.1 (9.16) | 67.2 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 29 | 21 | 24 | 19 | 28 | 18 | 14 | 208
  Male | 21 | 24 | 21 | 29 | 27 | 30 | 22 | 32 | 36 | 242
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  Asian-Central/South Asian Heritage | 0 | 0 | 4 | 0 | 3 | 1 | 2 | 2 | 3 | 15
  Asian-East Asian Heritage | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian-Japanese Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian-South East Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  White-Arabic/North African Heritage | 0 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 7
  White-White/Caucasian/European Heritage | 49 | 48 | 41 | 49 | 47 | 47 | 47 | 47 | 46 | 421

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 1-Primary Device Comparisons
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the health care practitioner (HCP) in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in patient instruction leaflets (PILs) for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in the primary DPI is presented. The analysis was performed on the Intent to Treat (ITT) Population which comprised of all enrolled participants who demonstrated use of their primary DPI.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | Symbicort Turbuhaler | Seretide Diskus | Spiriva Handihaler | Incruse/Anoro Ellipta | Ultibro/Seebri Breezhaler | Relvar Ellipta+LAMA | Symbicort Turbuhaler+LAMA | Seretide Diskus+LAMA
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 51 | 49 | 50 | 50 | 50
Percentage of participants | 10 | 40 | 26 | 34 | 10 | 33 | 12 | 38 | 26
Statistical Analysis 1: Comparison: Relvar Ellipta vs Symbicort Turbuhaler; Test type: Superiority; p = 0.005, Regression, Logistic — Analysis was performed using logistic regression with treatment cohort as fixed effect and adjusting for the covariate of time on current primary DPI; Odds Ratio (OR) = 4.657, 95% CI 2-sided [1.584 to 13.686] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta vs Seretide Diskus; Test type: Superiority; p = 0.114, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.478, 95% CI 2-sided [0.805 to 7.632] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 3: Comparison: Spiriva Handihaler vs Incruse/Anoro Ellipta; Test type: Superiority; p = 0.026, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.499, 95% CI 2-sided [1.160 to 10.555] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator
Statistical Analysis 4: Comparison: Incruse/Anoro Ellipta vs Ultibro/Seebri Breezhaler; Test type: Superiority; p = 0.012, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.943, 95% CI 2-sided [1.348 to 11.534] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator
Statistical Analysis 5: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.746, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.223, 95% CI 2-sided [0.361 to 4.151] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 6: Comparison: Relvar Ellipta vs Symbicort Turbuhaler; Test type: Superiority; p = 0.001, Regression, Logistic — Sensitivity analysis was performed using logistic regression with treatment cohort as fixed effect. Time on current primary device was removed from the model for this sensitivity analysis as it was confounded with primary device/treatment cohort; Odds Ratio (OR) = 5.562, 95% CI 2-sided [1.932 to 16.013] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 7: Comparison: Relvar Ellipta vs Seretide Diskus; Test type: Superiority; p = 0.050, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.979, 95% CI 2-sided [0.999 to 8.882] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 8: Comparison: Spiriva Handihaler vs Incruse/Anoro Ellipta; Test type: Superiority; p = 0.006, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 4.418, 95% CI 2-sided [1.521 to 12.834] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator
Statistical Analysis 9: Comparison: Incruse/Anoro Ellipta vs Ultibro/Seebri Breezhaler; Test type: Superiority; p = 0.009, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 4.165, 95% CI 2-sided [1.425 to 12.178] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator
Statistical Analysis 10: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.761, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 1.209, 95% CI 2-sided [0.357 to 4.095] — Odds ratio was calculated considering Relvar Ellipta as comparator

2. Primary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 1 in Primary DPI (Relvar Ellipta DPI Versus All ICS/LABA DPIs With a LAMA Second DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in the primary DPI is presented. The aim of the analysis was to compare percentage of participants making at least one critical error with Ellipta versus all ICS/LABA+LAMA DPIs; hence, the arms were combined as pre-specified in the protocol and reporting and analysis plan (RAP).
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Groups:
- [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]: All participants from Relvar Ellipta+LAMA, Symbicort Turbuhaler (Symb Turb)+LAMA, and Seretide Diskus+LAMA arms were included.
Arm/Group | [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] | Relvar Ellipta
Number analyzed (Participants) | 150 | 50
Percentage of participants | 25 | 10
Statistical Analysis 1: Comparison: [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] vs Relvar Ellipta; Test type: Superiority; p = 0.100, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.292, 95% CI 2-sided [0.853 to 6.163] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 2: Comparison: [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] vs Relvar Ellipta; Test type: Superiority; p = 0.051, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.642, 95% CI 2-sided [0.994 to 7.022] — Odds ratio was calculated considering Relvar Ellipta as comparator

3. Primary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 1 in Primary DPI (Relvar Ellipta With or Without a LAMA DPI) Versus Any Other ICS/LABA DPI With or Without a LAMA DPI
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in the primary DPI is presented. The aim of the analysis was to compare percentage of participants making at least one critical error with Ellipta and Ellipta+LAMA versus Turbuhaler and Turbuhaler+LAMA and Diskus and Diskus+LAMA; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Groups:
- Relvar Ellipta+[Relvar Ellipta+LAMA]: All participants from Relvar Ellipta and Relvar Ellipta+LAMA arms were included.
- Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]: All participants from Symbicort Turbuhaler and Symbicort Turbuhaler+LAMA arms were included.
- Seretide Diskus+[Seretide Diskus+LAMA]: All participants from Seretide Diskus and Seretide Diskus+LAMA arms were included.
Arm/Group | Relvar Ellipta+[Relvar Ellipta+LAMA] | Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA] | Seretide Diskus+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 100 | 100 | 100
Percentage of participants | 11 | 39 | 26
Statistical Analysis 1: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.995, 95% CI 2-sided [1.808 to 8.829] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.069, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.181, 95% CI 2-sided [0.940 to 5.059] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 3: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 4.855, 95% CI 2-sided [2.339 to 10.080] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 4: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.010, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.710, 95% CI 2-sided [1.274 to 5.764] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator

4. Primary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 1-Dual Device Comparisons (Relvar Ellipta DPI Versus Relvar Ellipta With Any Other LAMA)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in either one or both devices (where applicable) is presented.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | Relvar Ellipta+LAMA
Number analyzed (Participants) | 50 | 50
Percentage of participants | 10 | 22
Statistical Analysis 1: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.108, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.503, 95% CI 2-sided [0.818 to 7.659] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.122, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.409, 95% CI 2-sided [0.792 to 7.331] — Odds ratio was calculated considering Relvar Ellipta as comparator

5. Primary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 1-Dual Device Comparisons (Relvar Ellipta DPI Versus All ICS/LABA DPIs With a LAMA Second DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in either one or both devices (where applicable) is presented. The aim of the analysis was to compare percentage of participants making at least one critical error with Ellipta versus all ICS/LABA+LAMA DPIs; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 50 | 150
Percentage of participants | 10 | 41
Statistical Analysis 1: Comparison: Relvar Ellipta vs [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.887, 95% CI 2-sided [1.851 to 12.903] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta vs [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 5.484, 95% CI 2-sided [2.106 to 14.284] — Odds ratio was calculated considering Relvar Ellipta as comparator

6. Primary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 1-Dual Device Comparisons (Relvar Ellipta With or Without a LAMA DPI) Versus Any Other ICS/LABA DPI With or Without a LAMA DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in either one or both devices (where applicable) is presented. The aim of the analysis was to compare percentage of participants making at least one critical error with Ellipta and Ellipta+LAMA versus Turbuhaler and Turbuhaler+LAMA and Diskus and Diskus+LAMA; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta+[Relvar Ellipta+LAMA] | Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA] | Seretide Diskus+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 100 | 100 | 100
Percentage of participants | 16 | 47 | 36
Statistical Analysis 1: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.941, 95% CI 2-sided [1.863 to 8.337] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.030, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.391, 95% CI 2-sided [1.088 to 5.256] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 3: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 4.728, 95% CI 2-sided [2.388 to 9.364] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 4: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.957, 95% CI 2-sided [1.473 to 5.936] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator

7. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 1-Primary Device Comparisons
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. The percentage of participants with at least one overall error in the primary DPI is presented.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | Symbicort Turbuhaler | Seretide Diskus | Spiriva Handihaler | Incruse/Anoro Ellipta | Ultibro/Seebri Breezhaler | Relvar Ellipta+LAMA | Symbicort Turbuhaler+LAMA | Seretide Diskus+LAMA
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 51 | 49 | 50 | 50 | 50
Percentage of participants | 34 | 64 | 60 | 74 | 37 | 55 | 34 | 70 | 66
Statistical Analysis 1: Comparison: Relvar Ellipta vs Symbicort Turbuhaler; Test type: Superiority; p = 0.045, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.404, 95% CI 2-sided [1.018 to 5.676] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta vs Seretide Diskus; Test type: Superiority; p = 0.172, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.823, 95% CI 2-sided [0.770 to 4.319] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 3: Comparison: Spiriva Handihaler vs Incruse/Anoro Ellipta; Test type: Superiority; p = 0.016, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.989, 95% CI 2-sided [1.229 to 7.272] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator
Statistical Analysis 4: Comparison: Incruse/Anoro Ellipta vs Ultibro/Seebri Breezhaler; Test type: Superiority; p = 0.179, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.747, 95% CI 2-sided [0.775 to 3.937] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator
Statistical Analysis 5: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.690, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.189, 95% CI 2-sided [0.509 to 2.775] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 6: Comparison: Relvar Ellipta vs Symbicort Turbuhaler; Test type: Superiority; p = 0.004, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 3.363, 95% CI 2-sided [1.480 to 7.639] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 7: Comparison: Relvar Ellipta vs Seretide Diskus; Test type: Superiority; p = 0.012, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.848, 95% CI 2-sided [1.264 to 6.420] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 8: Comparison: Spiriva Handihaler vs Incruse/Anoro Ellipta; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 4.630, 95% CI 2-sided [1.986 to 10.791] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator
Statistical Analysis 9: Comparison: Incruse/Anoro Ellipta vs Ultibro/Seebri Breezhaler; Test type: Superiority; p = 0.081, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.037, 95% CI 2-sided [0.916 to 4.528] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator
Statistical Analysis 10: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 1.000, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.438 to 2.283] — Odds ratio was calculated considering Relvar Ellipta as comparator

8. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 1 in Primary DPI (Relvar Ellipta DPI Versus All ICS/LABA DPIs With a LAMA Second DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. The percentage of participants with at least one overall error in primary DPI is presented. The aim of the analysis was to compare percentage of participants making at least one overall error with Ellipta versus all ICS/LABA+LAMA DPIs; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] | Relvar Ellipta
Number analyzed (Participants) | 150 | 50
Percentage of participants | 57 | 34
Statistical Analysis 1: Comparison: [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] vs Relvar Ellipta; Test type: Superiority; p = 0.067, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.935, 95% CI 2-sided [0.955 to 3.921] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 2: Comparison: [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] vs Relvar Ellipta; Test type: Superiority; p = 0.007, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.523, 95% CI 2-sided [1.283 to 4.961] — Odds ratio was calculated considering Relvar Ellipta as comparator

9. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 1 in Primary DPI (Relvar Ellipta With or Without a LAMA DPI) Versus Any Other ICS/LABA DPI With or Without a LAMA DPI
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. The percentage of participants with at least one overall error in primary DPI is presented. The aim of the analysis was to compare percentage of participants making at least one overall error with Ellipta and Ellipta+LAMA versus Turbuhaler and Turbuhaler+LAMA and Diskus and Diskus+LAMA; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta+[Relvar Ellipta+LAMA] | Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA] | Seretide Diskus+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 100 | 100 | 100
Percentage of participants | 34 | 67 | 63
Statistical Analysis 1: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.008, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.399, 95% CI 2-sided [1.252 to 4.596] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.082, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.812, 95% CI 2-sided [0.926 to 3.544] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 3: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 3.840, 95% CI 2-sided [2.135 to 6.905] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 4: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 3.231, 95% CI 2-sided [1.810 to 5.766] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator

10. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 1-Dual Device Comparisons (Relvar Ellipta DPI Versus Relvar Ellipta With Any Other LAMA)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. The percentage of participants making at least one overall error in either one or both devices (where applicable) is presented.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | Relvar Ellipta+LAMA
Number analyzed (Participants) | 50 | 50
Percentage of participants | 34 | 46
Statistical Analysis 1: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.120, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.931, 95% CI 2-sided [0.842 to 4.428] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.232, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 1.636, 95% CI 2-sided [0.730 to 3.664] — Odds ratio was calculated considering Relvar Ellipta as comparator

11. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 1-Dual Device Comparisons (Relvar Ellipta DPI Versus All ICS/LABA DPIs With a LAMA Second DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. Errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. Percentage of participants making at least one overall error in either one or both devices (where applicable) is presented. The aim of the analysis was to compare percentage of participants making at least one overall error with Ellipta versus all ICS/LABA+LAMA DPIs; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 50 | 150
Percentage of participants | 34 | 71
Statistical Analysis 1: Comparison: Relvar Ellipta vs [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.217, 95% CI 2-sided [2.019 to 8.807] — Odds ratio was calculated considering Relvar Ellipta as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta vs [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 5.410, 95% CI 2-sided [2.660 to 11.005] — Odds ratio was calculated considering Relvar Ellipta as comparator

12. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 1-Dual Device Comparisons (Relvar Ellipta With or Without a LAMA DPI) Versus Any Other ICS/LABA DPI With or Without a LAMA DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. Errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. Percentage of participants making at least one overall error in either one or both devices (where applicable) is presented.The aim of the analysis was to compare percentage of participants making at least one overall error with Ellipta and Ellipta+LAMA versus Turbuhaler and Turbuhaler+LAMA and Diskus and Diskus+LAMA; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Day 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta+[Relvar Ellipta+LAMA] | Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA] | Seretide Diskus+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 100 | 100 | 100
Percentage of participants | 40 | 72 | 74
Statistical Analysis 1: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.007, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.477, 95% CI 2-sided [1.274 to 4.815] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 2: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.006, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.748, 95% CI 2-sided [1.328 to 5.683] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 3: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 3.896, 95% CI 2-sided [2.133 to 7.118] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator
Statistical Analysis 4: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 4.777, 95% CI 2-sided [2.508 to 9.100] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator

13. Secondary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 2-Primary Device Comparisons
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in the primary DPI is presented.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | Symbicort Turbuhaler | Seretide Diskus | Spiriva Handihaler | Incruse/Anoro Ellipta | Ultibro/Seebri Breezhaler | Relvar Ellipta+LAMA | Symbicort Turbuhaler+LAMA | Seretide Diskus+LAMA
Number analyzed (Participants) | 50 | 48 | 45 | 47 | 50 | 47 | 49 | 49 | 46
Percentage of participants | 0 | 8 | 11 | 21 | 0 | 17 | 6 | 6 | 13
Statistical Analysis 1: Comparison: Relvar Ellipta vs Symbicort Turbuhaler; Test type: Superiority; p = 0.176, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.347, 95% CI 2-sided [0.408 to 132.143] — Odds ratio was calculated considering Relvar Ellipta as comparator. Note: Statistical testing with a small number of events may produce unusual results; odds ratios and confidence intervals should be interpreted with caution
Statistical Analysis 2: Comparison: Relvar Ellipta vs Seretide Diskus; Test type: Superiority; p = 0.128, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 9.300, 95% CI 2-sided [0.526 to 164.465] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Spiriva Handihaler vs Incruse/Anoro Ellipta; Test type: Superiority; p = 0.038, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 20.454, 95% CI 2-sided [1.190 to 351.613] — Odds ratio was calculated considering Incruse/Anoro Ellipta as comparator. Note: Statistical testing with a small number of events may produce unusual results; odds ratios and confidence intervals should be interpreted with caution
Statistical Analysis 4: Comparison: Incruse/Anoro Ellipta vs Ultibro/Seebri Breezhaler; Test type: Superiority; p = 0.041, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 18.776, 95% CI 2-sided [1.131 to 311.669] — [estimate comment as in outcome 13, analysis 3]
Statistical Analysis 5: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.141, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 8.873, 95% CI 2-sided [0.484 to 162.775] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Relvar Ellipta vs Symbicort Turbuhaler; Test type: Superiority; p = 0.126, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 10.215, 95% CI 2-sided [0.519 to 200.904] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Relvar Ellipta vs Seretide Diskus; Test type: Superiority; p = 0.082, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 13.717, 95% CI 2-sided [0.715 to 263.125] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Spiriva Handihaler vs Incruse/Anoro Ellipta; Test type: Superiority; p = 0.024, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 28.283, 95% CI 2-sided [1.561 to 512.532] — [estimate comment as in outcome 13, analysis 3]
Statistical Analysis 9: Comparison: Incruse/Anoro Ellipta vs Ultibro/Seebri Breezhaler; Test type: Superiority; p = 0.038, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 21.736, 95% CI 2-sided [1.183 to 399.541] — [estimate comment as in outcome 13, analysis 3]
Statistical Analysis 10: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.188, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 7.603, 95% CI 2-sided [0.371 to 155.763] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 2 in Primary DPI (Relvar Ellipta DPI Versus All ICS/LABA DPIs With a LAMA Second DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in the primary DPI is presented. The aim of the analysis was to compare percentage of participants making at least one critical error with Ellipta versus all ICS/LABA+LAMA DPIs; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] | Relvar Ellipta
Number analyzed (Participants) | 144 | 50
Percentage of participants | 8 | 0
Statistical Analysis 1: Comparison: [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] vs Relvar Ellipta; Test type: Superiority; p = 0.147, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.781, 95% CI 2-sided [0.488 to 124.117] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] vs Relvar Ellipta; Test type: Superiority; p = 0.120, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 9.786, 95% CI 2-sided [0.553 to 173.301] — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 2 in Primary DPI (Relvar Ellipta With or Without a LAMA DPI) Versus Any Other ICS/LABA DPI With or Without a LAMA DPI
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in the primary DPI is presented. The aim of the analysis was to compare percentage of participants making at least one critical error with Ellipta and Ellipta+LAMA versus Turbuhaler and Turbuhaler+LAMA and Diskus and Diskus+LAMA; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta+[Relvar Ellipta+LAMA] | Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA] | Seretide Diskus+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 99 | 97 | 91
Percentage of participants | 3 | 7 | 12
Statistical Analysis 1: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.395, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.089, 95% CI 2-sided [0.383 to 11.389] — Odds ratio was calculated considering Relvar Ellipta+[Relvar Ellipta+LAMA] as comparator. Note: Statistical testing with a small number of events may produce unusual results; odds ratios and confidence intervals should be interpreted with caution
Statistical Analysis 2: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.166, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.250, 95% CI 2-sided [0.612 to 17.244] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.175, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 3.196, 95% CI 2-sided [0.596 to 17.140] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.042, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 5.408, 95% CI 2-sided [1.059 to 27.610] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 2-Dual Device Comparisons (Relvar Ellipta DPI Versus Relvar Ellipta With Any Other LAMA)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in either one or both devices (where applicable) is presented.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | Relvar Ellipta+LAMA
Number analyzed (Participants) | 50 | 49
Percentage of participants | 0 | 8
Statistical Analysis 1: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.090, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 12.145, 95% CI 2-sided [0.680 to 216.818] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.130, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 9.991, 95% CI 2-sided [0.508 to 196.435] — [estimate comment as in outcome 13, analysis 1]

17. Secondary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 2-Dual Device Comparisons (Relvar Ellipta DPI Versus All ICS/LABA DPIs With a LAMA Second DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in either one or both devices (where applicable) is presented. The aim of the analysis was to compare percentage of participants making at least one critical error with Ellipta versus all ICS/LABA+LAMA DPIs; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 50 | 144
Percentage of participants | 0 | 13
Statistical Analysis 1: Comparison: Relvar Ellipta vs [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.079, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 11.907, 95% CI 2-sided [0.753 to 188.208] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Relvar Ellipta vs [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.063, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 15.060, 95% CI 2-sided [0.866 to 262.042] — [estimate comment as in outcome 13, analysis 1]

18. Secondary Outcome: Percentage of Participants Making at Least One Critical Error at Visit 2-Dual Device Comparisons (Relvar Ellipta With or Without a LAMA DPI) Versus Any Other ICS/LABA DPI With or Without a LAMA DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose. The percentage of participants making at least one critical error in either one or both devices (where applicable) is presented. The aim of the analysis was to compare percentage of participants making at least one critical error with Ellipta and Ellipta+LAMA versus Turbuhaler and Turbuhaler+LAMA and Diskus and Diskus+LAMA; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta+[Relvar Ellipta+LAMA] | Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA] | Seretide Diskus+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 99 | 97 | 91
Percentage of participants | 4 | 11 | 13
Statistical Analysis 1: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.239, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.670, 95% CI 2-sided [0.521 to 13.690] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.200, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.929, 95% CI 2-sided [0.567 to 15.125] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.078, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 4.269, 95% CI 2-sided [0.848 to 21.489] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.046, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 5.132, 95% CI 2-sided [1.031 to 25.550] — [estimate comment as in outcome 15, analysis 1]

19. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 2-Primary Device Comparisons
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. The percentage of participants making at least one overall error in the primary DPI is presented.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | Symbicort Turbuhaler | Seretide Diskus | Spiriva Handihaler | Incruse/Anoro Ellipta | Ultibro/Seebri Breezhaler | Relvar Ellipta+LAMA | Symbicort Turbuhaler+LAMA | Seretide Diskus+LAMA
Number analyzed (Participants) | 50 | 48 | 45 | 47 | 50 | 47 | 49 | 49 | 46
Percentage of participants | 12 | 35 | 27 | 36 | 8 | 32 | 14 | 14 | 28
Statistical Analysis 1: Comparison: Relvar Ellipta vs Symbicort Turbuhaler; Test type: Superiority; p = 0.020, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.483, 95% CI 2-sided [1.218 to 9.961] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Relvar Ellipta vs Seretide Diskus; Test type: Superiority; p = 0.143, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.284, 95% CI 2-sided [0.757 to 6.895] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Spiriva Handihaler vs Incruse/Anoro Ellipta; Test type: Superiority; p = 0.006, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.268, 95% CI 2-sided [1.615 to 17.187] — [estimate comment as in outcome 13, analysis 3]
Statistical Analysis 4: Comparison: Incruse/Anoro Ellipta vs Ultibro/Seebri Breezhaler; Test type: Superiority; p = 0.009, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.655, 95% CI 2-sided [1.478 to 14.666] — [estimate comment as in outcome 13, analysis 3]
Statistical Analysis 5: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.679, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.274, 95% CI 2-sided [0.405 to 4.005] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Relvar Ellipta vs Symbicort Turbuhaler; Test type: Superiority; p = 0.010, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 3.804, 95% CI 2-sided [1.372 to 10.544] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Relvar Ellipta vs Seretide Diskus; Test type: Superiority; p = 0.083, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.555, 95% CI 2-sided [0.886 to 7.369] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Spiriva Handihaler vs Incruse/Anoro Ellipta; Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 5.930, 95% CI 2-sided [1.890 to 18.611] — [estimate comment as in outcome 13, analysis 3]
Statistical Analysis 9: Comparison: Incruse/Anoro Ellipta vs Ultibro/Seebri Breezhaler; Test type: Superiority; p = 0.007, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 4.929, 95% CI 2-sided [1.556 to 15.612] — [estimate comment as in outcome 13, analysis 3]
Statistical Analysis 10: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.746, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 1.208, 95% CI 2-sided [0.385 to 3.788] — [estimate comment as in outcome 13, analysis 1]

20. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 2 in Primary DPI (Relvar Ellipta DPI Versus All ICS/LABA DPIs With a LAMA Second DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps listed in PILs for the respective DPI. The errors were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per PIL. Overall errors is the combination of critical and non-critical errors. The percentage of participants making at least one overall error in primary DPI is presented. The aim of the analysis was to compare percentage of participants making at least one overall error with Ellipta versus all ICS/LABA+LAMA DPIs; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] | Relvar Ellipta
Number analyzed (Participants) | 144 | 50
Percentage of participants | 19 | 12
Statistical Analysis 1: Comparison: [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] vs Relvar Ellipta; Test type: Superiority; p = 0.404, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.502, 95% CI 2-sided [0.578 to 3.905] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA] vs Relvar Ellipta; Test type: Superiority; p = 0.330, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 1.591, 95% CI 2-sided [0.625 to 4.050] — [estimate comment as in outcome 13, analysis 1]

21. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 2 in Primary DPI (Relvar Ellipta With or Without a LAMA DPI) Versus Any Other ICS/LABA DPI With or Without a LAMA DPI
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps listed in PILs for the respective DPI. The errors were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per PIL. Overall errors is the combination of critical and non-critical errors. The percentage of participants making at least one overall error in primary DPI is presented. The aim of the analysis was to compare percentage of participants making at least one overall error with Ellipta and Ellipta+LAMA versus Turbuhaler and Turbuhaler+LAMA and Diskus and Diskus+LAMA; hence, the arms were combined as pre-specified in the protocol and RAP.
  .
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta+[Relvar Ellipta+LAMA] | Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA] | Seretide Diskus+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 99 | 97 | 91
Percentage of participants | 13 | 25 | 27
Statistical Analysis 1: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.189, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.738, 95% CI 2-sided [0.761 to 3.968] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.086, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.079, 95% CI 2-sided [0.901 to 4.799] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.082, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 1.950, 95% CI 2-sided [0.918 to 4.142] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.018, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.415, 95% CI 2-sided [1.161 to 5.024] — [estimate comment as in outcome 15, analysis 1]

22. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 2-Dual Device Comparisons (Relvar Ellipta DPI Versus Relvar Ellipta With Any Other LAMA)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. The percentage of participants making at least one overall error in either one or both devices (where applicable) is presented.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | Relvar Ellipta+LAMA
Number analyzed (Participants) | 50 | 49
Percentage of participants | 12 | 16
Statistical Analysis 1: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.472, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.510, 95% CI 2-sided [0.492 to 4.633] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Relvar Ellipta vs Relvar Ellipta+LAMA; Test type: Superiority; p = 0.553, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 1.402, 95% CI 2-sided [0.459 to 4.283] — [estimate comment as in outcome 13, analysis 1]

23. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 2-Dual Device Comparisons (Relvar Ellipta DPI Versus All ICS/LABA DPIs With a LAMA Second DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on correct use of inhalers. Any error made by the participant was recorded by HCP in the checklist. Checklist of instructions for correct use were based on steps for correct use listed in PILs for the respective DPI. Errors made during demonstration by participants were defined as critical, when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per PIL. Overall errors is the combination of critical and non-critical errors. Percentage of participants making at least one overall error in either one or both devices (where applicable) is presented. The aim of the analysis was to compare percentage of participants making at least one overall error with Ellipta versus all ICS/LABA+LAMA DPIs; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta | [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 50 | 144
Percentage of participants | 12 | 29
Statistical Analysis 1: Comparison: Relvar Ellipta vs [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.052, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.523, 95% CI 2-sided [0.993 to 6.407] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Relvar Ellipta vs [Relvar Ellipta+LAMA]+[Symb Turb+LAMA]+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.029, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.757, 95% CI 2-sided [1.107 to 6.862] — [estimate comment as in outcome 13, analysis 1]

24. Secondary Outcome: Percentage of Participants Making at Least One Overall Error at Visit 2-Dual Device Comparisons (Relvar Ellipta With or Without a LAMA DPI) Versus Any Other ICS/LABA DPI With or Without a LAMA DPI)
Description: Participants were asked to demonstrate use of their prescribed DPI at Visit 2 within 6 weeks after they were retrained on the correct use of inhalers. Any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical", when the participant received a lesser/no dose and non-critical when the dose may not be affected, but the participant has demonstrated improper use of their DPI, as per the PIL. Overall errors is the combination of critical and non-critical errors. The aim of the analysis was to compare percentage of participants making at least one overall error with Ellipta and Ellipta+LAMA versus Turbuhaler and Turbuhaler+LAMA and Diskus and Diskus+LAMA; hence, the arms were combined as pre-specified in the protocol and RAP.
Time Frame: Week 6
Population: ITT Population. Only those participants with data available at Visit 2 were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Relvar Ellipta+[Relvar Ellipta+LAMA] | Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA] | Seretide Diskus+[Seretide Diskus+LAMA]
Number analyzed (Participants) | 99 | 97 | 91
Percentage of participants | 14 | 33 | 34
Statistical Analysis 1: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.024, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.434, 95% CI 2-sided [1.123 to 5.276] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.035, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.389, 95% CI 2-sided [1.061 to 5.376] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Symbicort Turbuhaler+[Symbicort Turbuhaler+LAMA]; Test type: Superiority; p = 0.003, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.889, 95% CI 2-sided [1.434 to 5.819] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: Relvar Ellipta+[Relvar Ellipta+LAMA] vs Seretide Diskus+[Seretide Diskus+LAMA]; Test type: Superiority; p = 0.003, Regression, Logistic — [p-value comment as in outcome 1, analysis 6]; Odds Ratio (OR) = 2.974, 95% CI 2-sided [1.461 to 6.055] — [estimate comment as in outcome 15, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected until completion of the study (Up to Week 6)
Description: SAEs and non-SAEs were collected in the ITT Population.
Arm/Group | Relvar Ellipta | Symbicort Turbuhaler | Seretide Diskus | Spiriva Handihaler | Incruse/Anoro Ellipta | Ultibro/Seebri Breezhaler | Relvar Ellipta+LAMA | Symbicort Turbuhaler+LAMA | Seretide Diskus+LAMA
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50 | 0/51 | 0/49 | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50 | 1/51 | 1/49 | 0/50 | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 4/50 | 1/50 | 0/50 | 1/50 | 2/51 | 2/49 | 3/50 | 3/50 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relvar Ellipta (N=50) | Symbicort Turbuhaler (N=50) | Seretide Diskus (N=50) | Spiriva Handihaler (N=50) | Incruse/Anoro Ellipta (N=51) | Ultibro/Seebri Breezhaler (N=49) | Relvar Ellipta+LAMA (N=50) | Symbicort Turbuhaler+LAMA (N=50) | Seretide Diskus+LAMA (N=50)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relvar Ellipta (N=50) | Symbicort Turbuhaler (N=50) | Seretide Diskus (N=50) | Spiriva Handihaler (N=50) | Incruse/Anoro Ellipta (N=51) | Ultibro/Seebri Breezhaler (N=49) | Relvar Ellipta+LAMA (N=50) | Symbicort Turbuhaler+LAMA (N=50) | Seretide Diskus+LAMA (N=50)
Chronic obstructive (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 3 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT03114969/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT03114969/SAP_001.pdf